CLINICAL TRIAL: NCT02635230
Title: An International Prospective Registry on Concomitant Use of Oral Anticoagulants and P2Y12 Inhibitors in Patients With Atrial Fibrillation or Heart Valve Prosthesis Undergoing Coronary Revascularisation.
Brief Title: What is the Optimal antiplatElet and Anticoagulant Therapy in Patients With Oral Anticoagulation Undergoing revasculariSaTion 2.
Acronym: WOEST 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: R&D Cardiologie (Other)
Collaborators: St. Antonius Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R&D/Z14.016/WOEST2; WOEST2-004 (Other: WOEST 2 Study Team); V.21483/W14.007 (Other: Medical research Ethics Committees United - St. Antonius Hospital, the Netherlands)
Record Dates: First submitted 2015-12-10; First posted 2015-12-18 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillations; Heart Valve Prostheses; Acute Coronary Syndromes; Coronary Artery Diseases; Stroke; Bleeding; Myocardial Infarction
Keywords: Atrial Fibrillations; Heart Valve Prostheses; Acute Coronary Syndromes; Percutaneous Coronary Revascularization; Coronary Artery Bypass Grafting; Coronary Artery Diseases; Myocardial Infarction; Ischemic stroke; Bleeding; Thrombosis; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Embolism and Thrombosis; Platelet Aggregation Inhibitors; Aspirin; Clopidogrel; Ticagrelor; Prasugrel; Antithrombotic treatment; Oral anticoagulation; Warfarin; Dabigatran etexilate mesylate; Apixaban; Rivaroxaban; Direct Factor Xa Inhibitors; Direct Thrombin Inhibitors
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome; Coronary Artery Disease; Stroke; Hemorrhage; Myocardial Infarction; Ischemic Stroke; Thrombosis; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Embolism and Thrombosis | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic oral anticoagulation and P2Y12 inhibitor: Patients with chronic indication for chronic oral anticoagulation (OAC) because of a heart valve prosthesis and/or atrial fibrillation undergoing coronary revascularisation (by PCI or CABG) and requiring concomitant treatment with P2Y12 inhibitors.
  Interventions: Drug: Combination of chronic oral anticoagulation and a P2Y12 inhibitor with or without aspirin.

INTERVENTIONS:
Drug: Combination of chronic oral anticoagulation and a P2Y12 inhibitor with or without aspirin.

SUMMARY:
The optimal antithrombotic therapy for patients with atrial fibrillation (AF) with a CHA2DS2-VASc score ≥1 with concomitant acute coronary syndrome (ACS) or revascularisation by percutaneous coronary intervention (PCI) with stenting, is still unknown. For these patients current North American and European guidelines recommend a triple therapy strategy, including vitamin K antagonists (VKA), aspirin and clopidogrel. A major drawback of this triple therapy strategy is a significant increase in the risk of major bleeding. Furthermore, the ommitance of aspirin and the introduction of more potent P2Y12 inhibitors as well as the non-vitamin K oral anticoagulants (NOAC), created numerous new antithrombotic treatment strategies for these patients with overlapping conditions. To date, evidence on the risks and benefits of these new antithrombotic treatment strategies is lacking.

The WOEST 2 Registry aims to improve medical care for patients with AF and/or a heart valve prosthesis ánd undergoing coronary revascularisation through a better understanding of their demographics, antithrombotic management and related in-hospital and long-term outcomes. The WOEST 2 Registry will provide data to support benchmarking of antithrombotic treatment patterns and patient outcomes.

Objective: To assess the different management patterns and related in-hospital and long-term safety and efficacy outcomes of combined use of chronic oral anticoagulation and a P2Y12 inhibitor in patients with atrial fibrillation and/or a heart valve prosthesis undergoing coronary revascularisation.

DETAILED DESCRIPTION:
The WOEST 2 Registry is a prospective, international, multi-centre, non-interventional, cohort study designed to recruit an unselected cohort of patients with atrial fibrillation and/or a heart valve prosthesis undergoing coronary revascularisation.

Trial overview

Name : WOEST 2 REGISTRY

Target for enrollment : 2200 patients

Time frame for inclusion : within 72 hours after index PCI or coronary artery bypass grafting (CABG)

Follow-up : 24 months

Visits : 30 days, 12 and 24 months after index PCI or CABG

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to be included in this registry, a subject must meet ALL of the following criteria:

1. Patient is ≥ 18 years of age;
2. Patients with a diagnosis of atrial fibrillation (prior to hospitalisation ór during hospitalisation within 72h after coronary revascularisation) and/or with a heart valve prosthesis (aortic/mitral);
3. Chronic treatment with OAC or NOAC therapy at inclusion or the intention to start chronic treatment with OAC or NOAC within 72h after coronary revascularisation AND with intended duration of treatment for at least one year after inclusion in the registry;
4. Indication for coronary revascularisation by CABG or PCI (with deployment of at least 1 coronary stent);
5. Prescription of a P2Y12 inhibitor (clopidogrel, ticagrelor or prasugrel) because of CABG following acute coronary syndrome* and /or because of PCI (with deployment of at least 1 coronary stent).
6. Patient has provided written informed consent.

Exclusion Criteria:

A potential subject who meets ANY of the following criteria will be excluded from participation in this study:

1. Patients unable to sign informed consent (including mental disabled patients);
2. Patients with life expectancy < 1 year;
3. Allergy or intolerance to P2Y12 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: WOEST2 Registry is designed to recruit an unselected cohort of patients with AF and/or a heart valve prosthesis undergoing coronary revascularisation (PCI/CABG) within at least three European countries (Netherlands, Belgium, United Kingdom). The three international cohorts of patients reflect the spectrum of our study population within the geographic catchment regions. At least 15 hospitals of varying size and characteristics will participate in this study.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2014-06; Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Composite of the rate of non-fatal myocardial infarction, non-fatal ischemic stroke (including transient ischemic attack), non-central nervous system systemic embolization and cardiovascular death [the primary efficacy outcome]. | 1 year
The occurrence of any bleeding episode requiring in-hospital medical attention and/or a switch of antithrombotic medication [the primary safety outcome]. | 1 year
  Bleeding will be classified by the Bleeding Academic Research Consortium (BARC) 2, 3, 4 and 5 bleeding criteria and by the Thrombolysis in Myocardial Infarction (TIMI) minor and major bleeding criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jurriën M ten Berg, MD, PhD, Principal Investigator — St. Antonius Hospital Nieuwegein, the Netherlands; Willem JM Dewilde, MD, PhD, Principal Investigator — Imelda Hospital Bonheiden, Belgium
Locations (9):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis Leuven, Leuven
- Netherlands (4):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amphia Ziekenhuis, Breda
  - St. Antonius Hospital, Nieuwegein
  - Elizabeth-TweeSteden Ziekenhuis, Tilburg